CLINICAL TRIAL: NCT00391833
Title: Effect of Panax Ginseng on the Cognitive Performance in Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ginseng-AD
Record Dates: First submitted 2006-10-22; First posted 2006-10-24 (Estimated); Last update posted 2006-10-24 (Estimated); Status verified 2006-10

CONDITIONS: Alzheimer's Disease; Memory Decline
Keywords: Alzheimer's disease, Ginseng, CD34
MeSH Terms: conditions — Alzheimer Disease | interventions — Asian ginseng

INTERVENTIONS:
Drug: Panax Ginseng

SUMMARY:
We investigate the clinical efficacy of Panax ginseng in Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is characterized by a progressive decline of memory and intellectual abilities, interfering activity in daily living, the overall quality of life, and ultimately leads to death. Although pharmacologic treatments are currently approved for treating mild- to moderate AD using acetylcholinesterase inhibitors (ACEI) or memantine, the NMDA antagonist, for the advanced stage of AD, the therapeutic efficacies need to be further improved.

For millennia, ginseng or its components have been used to treat medical conditions, and the pharmacologic effects have been demonstrated in cardiovascular, endocrine and immune system (Attele et al., 1999). In means of memory and learning, a number of studies suggested that ginseng can attenuate learning deficits of damaged or ageing brains in rodent models (Kennedy et al., 2003; Zhao and McDaniel, 1998; Nitta et al., 1995). In studies with human healthy participants, correspondently, both acute and chronic dosage of ginseng increased the cognitive performance (Kennedy et al., 2001; Kennedy et al., 2003; D'Angelo et al., 1986; Sorensen and Sonne, 1996).

In this study, we we will investigate the contribution of ginseng treatment in increasing the cognitive improvement of AD patients. In addition, we will test various bio-markers and hematopoietic progenitor cell count in those included patients using their blood samples. Patients with AD as well as memory decline will be included

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease

Exclusion Criteria:

* other neurologic disease

Ages: 40 Years to 83 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2004-04; Study Completion 2005-10

PRIMARY OUTCOMES:
Cognitive performances monitored by MMSE and Alzheimer's disease assessment scales.
Biomarkers including hematopoietic progenitor cell count.

CONTACTS AND LOCATIONS:
Overall Officials: Manho Kim, MD, PhD, Study Chair — Department of Neurology, Seoul National University Hospital

REFERENCES:
- [Derived] Lee ST, Chu K, Sim JY, Heo JH, Kim M. Panax ginseng enhances cognitive performance in Alzheimer disease. Alzheimer Dis Assoc Disord. 2008 Jul-Sep;22(3):222-6. doi: 10.1097/WAD.0b013e31816c92e6. PMID 18580589